CLINICAL TRIAL: NCT07123948
Title: The Correlation Between Packed Red Blood Cell Transfusion and Early and Late Complications of Prematurity
Brief Title: The Correlation Between Red Cell Transfusion and Complications of Prematurity
Status: Not yet recruiting | Type: Observational
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Kristina Lah Tomulić, assoc. professor, Clinical Hospital Center Rijeka
Other Study IDs: 003-05/24-01/150
Record Dates: First submitted 2025-07-15; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Retinopathy of Prematurity (ROP); Bronchopulmonary Dysplasia (BPD); Enterocolitis, Necrotizing; Intraventricular Hemorrhage Neonatal
Keywords: Infant, Premature;; Erythrocyte Transfusion; Neurodevelopmental Disorder
MeSH Terms: conditions — Retinopathy of Prematurity; Bronchopulmonary Dysplasia; Enterocolitis, Necrotizing; Premature Birth; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assesment of the neurological and neurodevelopmental outcome at the age of six: All premature infants (less than 32 weeks of gestation) will be neurologically assessed at the age of six. Also, their neurodevelopmental outcome will be assessed at the age of six using the Wechsler Intelligence Test.
  Interventions: Diagnostic Test: Wechsler Intelligence Test, performed by educated psychologists

INTERVENTIONS:
Diagnostic Test: Wechsler Intelligence Test, performed by educated psychologists — At the age of six, parents of children who meet the inclusion criteria will receive a notification about the study from the responsible paediatrician. If they agree to participate, they will sign an informed consent form. They will then be invited to the clinic for a neurological and neurodevelopmental assessment. The neurological examination will be conducted by the principal investigator or collaborators who are paediatric specialists. The neurodevelopmental evaluation will be performed by a qualified psychologist using the Wechsler Intelligence Test.
  The Wechsler Intelligence Test for Children - Fourth Edition is a clinical tool for measuring the intelligence of children aged 6 to 16 years and 11 months. It assists in identifying specific learning difficulties, hyperactivity disorder, speech and language challenges, and intellectual impairments. The test comprises 15 subtests.

SUMMARY:
The aim of this clinical trial is to learn if there is a correlation between the erythrocyte transfusion in the early neonatal period in premature infants and early and late complications of prematurity. The main questions it aims to answer are:

* Do premature infants who receive blood transfusions within their first month of life have a higher risk of early prematurity complications, such as retinopathy of prematurity, necrotising enterocolitis, bronchopulmonary dysplasia, and intraventricular haemorrhage?
* Do premature infants who receive blood transfusions during their first month of life have worse neurological and neurodevelopmental outcomes than those who do not? The first part of the study is retrospective, using data collected from participants' histories. The second part is prospective, evaluating neurological and neurodevelopmental outcomes at the age of six years.

DETAILED DESCRIPTION:
Premature infants are the group that receives the most red blood cell transfusions. Between 50% and 90% of very low birth weight (VLBW) infants (less than 1500 g) and up to 95% of extremely low birth weight (ELBW) infants (less than 1000 g) will receive at least one red blood cell transfusion during hospitalisation.

To date, there are no clear guidelines for transfusion in premature infants in clinical practice.

Premature infants are particularly susceptible to tissue injury caused by impaired oxygen delivery, and complications are associated with this imbalance in tissue oxygenation. The pathophysiology of complications in transfused premature infants involves several interconnected mechanisms arising from organ immaturity and the specific effects of transfusion.

Over the past twenty years, numerous scientific studies have investigated the adverse effects of packed red blood cell transfusions. Many of these studies have associated red blood cell transfusions with a higher risk of both early and late complications of prematurity, such as necrotising enterocolitis (NEC), retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), intraventricular haemorrhage (IVH), and issues in later neurodevelopment. Only a few studies have reported beneficial effects of transfusion.

Red blood cell transfusion, along with other comorbidities in preterm infants, may contribute to neurological and neurodevelopmental damage. Some studies have confirmed that a restrictive approach leads to better neurodevelopmental outcomes, while others have shown abnormal brain structures and volumes at school age.

Based on previous research and the varied results obtained, the investigators aim to investigate the relationship between packed red blood cell transfusion, the number of transfusions, and the age at the time of transfusion concerning the occurrence of early and late prematurity complications. The investigators also seek to determine whether the haemoglobin level at the time of transfusion influences the development of complications. Although the impact on neurodevelopmental outcomes is partly understood and studied in younger premature children (aged 2 to 5), there are few studies and limited research on the effects in older children.

The hypothesis of this study is that premature infants who received packed red blood cell transfusions during the neonatal period have a higher rate of early prematurity complications and poorer neurological and neurodevelopmental outcomes at six years of age compared to premature infants who did not receive transfusions.

Investigation plan In the first, retrospective part, the investigators will collect epidemiological data from premature newborns (less then 32 weeks of gestation) from the hospital information system (IBIS) and the medical histories of the participants between June 2018 and December 2021.

The participants will be split into those who received a transfusion of packed red blood cells and those who did not.

In the second phase of the study, the investigators will evaluate the neurological and neurodevelopmental outcomes of the same participants during preschool age (at 6 years old adjusted for chronological age), based on the transfusion treatment. This phase will take place from September 2025 to December 2028. Parents of each child meeting the inclusion criteria will receive a notice about the study, which will be delivered by a primary care paediatrician during the examination that all children should have before starting their first year of primary school. After reading the notice, parents will sign the inform consent form if they agree to participate. The primary paediatrician will inform the main investigator, after which the child and parent or guardian will be invited to the Paediatrics Clinic for a neurological and neurodevelopmental assessment. Once all data collection is complete, statistical analysis will be performed to explore whether there is a connection between transfused preterm infants, early prematurity complications, and neurological and neurodevelopmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all children born as premature infants <32. weeks of gestation in Clinical Hospital Centre Rijeka from June 2018. to December 2021. (and who will be on September 2025. six years old)
* signed informed consent

Exclusion Criteria:

* genetic syndromes, severe congenital anomalies

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The participants will be identified and selected by the primary care paediatricians in Primorsko-Goranska, Istarska, and Ličko-Senjska County (western part of Croatia)
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Motor function at the age of 6 years in premature infants who received erythrocyte transfusion compared to those who did not | From enrollment to the end of the neurologic assessment at 4 weeks.
  The outcome measure is the motor function of premature infants (less than 32 weeks of gestation) at the age of 6 years who received erythrocyte transfusion in the neonatal period.
  The aim is to identify the proportion of participants with normal, mildly impaired, moderately impaired, or severely impaired motor function.
  The Gross Motor Function Classification System (GMFCS) will be used to assess motor function.
  GMFCS is a standardized classification tool used to evaluate and describe motor function levels in children with cerebral palsy. It was created to offer a dependable framework for understanding restrictions in gross motor skills in children of different age groups.
  If The GMFCS score is 0, motor function is normal. Cerebral palsy will be classified as mild if the GMFCS score is 1, moderate if the GMFCS score is 2, and severe if the GMFCS score is 3 or higher.
  On the GMFCS scale, the minimum value is 0, and the maximum value is 5. The higher score means a worse outcome.
Hearing assessment at the age of 6 years in premature infants who received erythrocyte transfusion compared to those who did not | From enrollment to the end of the hearing assessment at 4 weeks.
  The aim is to identify the proportion of participants with normal and impaired hearing function.
  Hearing assessment depends on whether the child requires hearing aids. If the child needs hearing aids, the score will be 1; if not, the score will be 0.
  The minimum value is 0, and the maximum value is 1. A higher score means a worse outcome.
Visual assessment at the age of 6 years in premature infants who received erythrocyte transfusion compared to those who did not | From enrollment to the end of the hearing assessment at 4 weeks.
  The aim is to identify the proportion of participants with normal and impaired visual function.
  Visual assessment depends on whether the child requires visual aids. If the child needs visual aids, the score will be 1; if not, the score will be 0.
  The minimum value is 0, and the maximum value is 1. A higher score means a worse outcome.
Neurodevelopmental outcome of premature infants who received erythrocyte transfusion compared to those who did not | From enrollment to the end of the neurologic assessment at 4 weeks.
  Neurodevelopmental assessment will be conducted using the Wechsler Intelligence Scale for Children (WISC-IV). It is a clinical tool for evaluating the intelligence of children aged 6 to 16 years and 11 months.
  The test includes 15 subtests - 10 core and 5 supplementary. Intellectual functioning in specific cognitive areas is also represented by four composite scores: the Verbal Comprehension Index (VCI), the Perceptual Reasoning Index (PRI), the Working Memory Index (WMI), and the Information Processing Speed Index (PSI). The total test score (UIQ) is calculated based on the sum of scaled scores across the 10 core subtests. The resulting IQ scores are categorized as follows: 69 and below is extremely low; 70 to 79 is borderline; 80 to 89 is low average; 90 to 109 is average; 110 to 119 is high average; 120 to 129 is superior; and 130 and above is very superior.
  Minimum value is 40, and the maximum value is 200. The higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: senada šerifi, Principal Investigator — Clinical Hospital Centre Rijeka, Croatia
Locations (1):
- Clinical Hospital Centre Rijeka, Department of Paediatrics, Rijeka, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: No
The ethics committee's initial decision was that the IPD would not be shared. However, the investigators may share the summarised and statistically processed data of the participants.